CLINICAL TRIAL: NCT06289010
Title: Neural Mechanisms of Evidence-Based, Family-Focused Treatment for Youth Depression: Preliminary Open Trial
Brief Title: Neural Mechanisms of Family-Focused Treatment for Youth Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7354E
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Childhood Depression
Keywords: Neural Mechanisms; Depression; Children; Adolescent; Family
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Depressed Group (Experimental): 20 children with depression and their parents (40 participants total) will undergo a 12-session course of FFT-CD.
  Interventions: Behavioral: Family-Focused Treatment for Childhood-Depression (FFT-CD)

INTERVENTIONS:
Behavioral: Family-Focused Treatment for Childhood-Depression (FFT-CD) — This intervention includes 12 one-hour, in-person sessions. FFT-CD was designed to help families gain skills to combat depression and create ways of interacting that protect the child from the negative sequelae of stress. Within a broad psychoeducational framework, interpersonal factors impacting youth depression and the interplay of mood and interpersonal interactions are emphasized. Participants are taught to identify Upward Spirals - positive interactions fueling positive moods leading further upward - and Downward Spirals - negative interactions fueling negative moods leading further downward. The treatment rationale is "to stop downward spirals and to start upward spirals"; this idea provides a foundation for skills building to help the child and family better navigate stress. Handouts, role-playing, behavioral rehearsal, and homework assignments are all used to help shape behaviors.

SUMMARY:
The goal of this interventional study is to compare the baseline neural mechanisms and parenting in depressed and non-depressed children and to examine baseline neural mechanisms and parenting as predictors of Family-Focused Treatment for Childhood-Depression (FFT-CD) outcomes. The main questions it aims to answer are:

* What are differences between depressed and non-depressed participants on baseline neural and parenting indicators?
* Do baseline neural and parenting indicators predict response to FFT-CD?
* Does change in parenting and neural functioning mediate change in depression from baseline to follow-up?

Participants will:

* complete baseline clinical measures
* complete neuroimaging tasks via Functional Magnetic Resonance Imaging (fMR)
* undergo a 12-session course of FFT-CD
* complete follow up evaluations and neuroimaging

DETAILED DESCRIPTION:
Childhood-onset depression is impairing, often recurrent and persistent, and negatively impacts development, resulting in high personal, social, and economic costs. Family-Focused Treatment for Childhood-Depression (FFT-CD) was developed to address the needs of depressed youth. In a large, randomized controlled trial, FFT-CD was superior to individual therapy in promoting recovery from depression.

Despite its promise, there was high variability in degree of improvement in FFT-CD. Our long-term goal is to integrate parenting, neuroimaging and clinical measures to a) reveal the parenting, emotional and neural mechanisms of clinical benefit for FFT-CD and (b) examine what parent and child characteristics predict immediate and long-term benefit. The proposed study will provide groundwork for this larger study by providing preliminary data.

This study will enroll 40 children (ages 7-12) - 20 with current depressive disorder and 20 with no history of mental health disorder -- and their parents (40 parents total). At baseline parents and children will participate in (a) an evaluation of clinical state and family functioning, (b) functional neuroimaging procedures to evaluate neural response to emotional cues (faces), potential reward, and parent-child relations, and resting state-connectivity, and (c) structural imaging (MRI and diffusion tensor imaging). Participants with depressive disorders and their parents will then be provided a 12-session course of FFT-CD. Brief clinical and parenting data will be collected at two points during treatment; baseline procedures will be repeated at 4 months (post-treatment). The participants will engage in briefer clinical evaluation via telehealth 6 and 9 months post-treatment.

Goals include: 1) To examine differences between depressed and non-depressed participants in baseline neural and parenting. 2) To examine baseline neural functioning, emotional experience, and parenting as predictors of FFT-CD outcome in our depressed group. 3) To evaluate parenting and emotional experience across treatment and neural functioning measures at the end of treatment as mediators of change in depression from baseline to final follow-up.

The neuroimaging hypotheses include:

* Naturalistic Videos Task: Children with depression will display greater amygdala and insula activation to negatively vs. neutrally valenced video clips. There will be less striatal activation to positively vs. neutrally valenced video clips in the depressed group compared to the n on-depressed group. Dyads of depressed children and their parents will show less functional similarity while viewing naturalistic clips of parent-child interactions compared to healthy control dyads.
* Face Matching Task: Depressed children will show amygdala and insula hyperactivation in response to negative faces and striatum hypoactivation in response to positive faces compared to healthy controls.
* Reward Processing Task: Depressed children will show reduced striatal activation in response to reward anticipation and receipt relative to healthy controls.
* Evaluative Comments Task: Depressed children will display higher activation in the default mode network during self-evaluation relative to non-depressed control children across both conditions. We further expect a greater heightened Default Mode Network (DMN) response in the depressed group to negative words relative to positive words.
* Rest: Dyads of depressed children and their parents will show less functional similarity in the resting state functional connectome relative to non-depressed control dyads. Greater DMN connectivity will be observed at rest in depressed children relative to non-depressed control children.
* Magnetic Resonance Spectroscopy: Depressed children will show elevated levels of glutamate, aspartate, choline, and lactate and lower levels of ascorbate, glutathione, myo-inositol, and N-acetyl aspartate relative to non-depressed controls, consistent with neuroinflammation and excitotoxicity/oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Children must:

  * Have a current DSM-5 diagnosis of MDD, Persistent DD, or DDNOS (based on K-SADS-PL) OR not meet criteria for any DSM-5 mental health diagnosis (based on K-SADS-PL)
  * Be ages 7-12
  * Be living with a parent(s) or guardian willing to participate
  * Be able and willing to provide informed consent/assent

Parent must:

* Not be currently pregnant
* Be able to read, understand consent forms, and provide consent on their child's behalf
* Be the biological parent (or grandparent in parental role) of the participating child & have lived with the child for more than 75% of the child's life.

All participants must:

* Not have a disturbance that would interfere with participation such as autism spectrum disorder, psychosis, current substance dependence, current use of psychotropic medication, OCD, or MRI contraindication such as metal inside the body or claustrophobia
* Be proficient in English

Exclusion Criteria:

* Thought or other disturbance in the child that would interfere with the ability to participate in treatment or assessments (e.g., psychotic disorder, autism spectrum disorder, OCD, active substance abuse/dependence, intellectual disability, as assessed on KSADS-PL)
* Severe conduct disorders in the child that threaten the home stability (e.g. juvenile justice or children's protective service involvement as assessed on KSADS-PL) due to the potential impact on retention
* Youth or primary caregivers do not speak English
* Either parent or child has contraindications for neuroimaging (e.g., claustrophobia, metal implants, braces, electronically, magnetically, or mechanically activated devices such as cochlear implants)
* The child is on an antidepressant medication, as it may complicate neuroimaging interpretation.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Depression Treatment Response | 4 months (post-treatment)
  >/= 50% reduction on Children's Depression Rating Scale-Revised (CDRS-R). Scores on this measure range from 17 to 113, and higher scores indicate greater depression severity.
Children's Self Report of Depressive Symptoms | 4 months
  Children's Depression Inventory (CDI) is a 28-item self-report measure. Scores range from 0 to 54 with higher scores reflecting higher levels of symptoms.

SECONDARY OUTCOMES:
Depression Remission | 4 months
  </= 28 score on Children's Depression Rating Scale-Revised (CDRS-R)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Boston University, Boston, Massachusetts
  - Athinoula A. Martinos Imaging Center at Massachusetts Institute of Technology, Charlestown, Massachusetts

IPD SHARING:
Plan to Share IPD: No
These are initial pilot data and will not be shared at this time.